CLINICAL TRIAL: NCT01429844
Title: Randomized, Open-label, Multi-Center Study Comparing Tacrolimus With Cyclosporin, Both Arms in Combination With Mycophenolate Mofetil and Corticosteroids for Prevention of Bronchiolitis Obliterans Syndrome in Lung Transplant Patients
Brief Title: Tacrolimus Versus Cyclosporine for Immunosuppression After Lung Transplantation
Acronym: EAILTX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hermann Reichenspurner, Prof. Dr. med. Hermann Reichenspurner, PhD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EAILTx Tac vs. CsA in LuTx
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Bronchiolitis Obliterans; Immunosuppression
Keywords: Calcineurin inhibitors; Bronchiolitis obliterans; Lung transplantation; Cyclosporine; Tacrolimus; Mycophenolate; Steroids; Chronic rejection; Acute rejection; Obliterative bronchiolitis
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus (Active Comparator): Tacrolimus in combination with mycophenolate mofetil and steroids for denovo immunosuppression after lung transplantation
  Interventions: Drug: Tacrolimus
- Cyclosporine (Active Comparator): Cyclopsorine in combination with mycophenolate mofetil and steroids for denovo immunosuppression after lung transplantation
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus therapy was started immediately after transplantation with a continuous intravenous infusion of 0.01-0.03 mg/kg/d. After extubation, the mode of delivery was switched to oral administration (b.i.d.) with doses of 0.05-0.3 mg/kg/d. Tacrolimus doses were adjusted to trough levels. Target C0 (trough) levels were 10-15 ng/ml for the first 3 months after transplantation and 8-12 ng/ml thereafter with dose adjustments according to patient outcome.
  Other Names: FK 506; Prograf
  Arms: Tacrolimus
Drug: Cyclosporine — Cyclosporine therapy was started immediately after transplantation with a continuous intravenous infusion of 1-3 mg/kg/d. After extubation the mode of delivery was switched to oral administration (b.i.d. or t.i.d.) with doses of 4-18 mg/kg/d. Cyclosporine doses were adjusted to C0 or C2 levels according to local practice. Target trough levels were 200 - 300 ng/ml for the first 3 months after transplantation and 150 - 200 ng/ml thereafter.
  Other Names: CyA; CsA; Cyclosporine A; Sandimmune
  Arms: Cyclosporine

SUMMARY:
The purpose of the study is to compare efficacy and safety of two different immunosuppressive regimens for prevention of bronchiolitis obliterans syndrome (BOS) (chronic lung allograft rejection)after lung transplantation: tacrolimus versus cyclosporine, both in combination with mycophenolate mofetil and steroids. The study was powered to detect a 15% reduction in BOS in tacrolimus treated patients.

Study design: open-label, randomized, comparative, multi-center, investigator driven

DETAILED DESCRIPTION:
Lung transplantation has become a viable treatment option for selected patients with end stage lung disease and leads to prolonged survival and improved quality of life. However, despite improvements in surgical techniques, immunosuppressive therapies and long-term care, survival rates reported by the Registry of the International Society for Heart and Lung Transplantation (ISHLT) (79% 1-year and 52% 5-year) are lower than those reported for other solid organ transplants. The leading cause of death in long-term follow-up after lung transplantation is chronic allograft dysfunction due to obliterative bronchiolitis (OB) manifested by its physiological correlate the bronchiolitis obliterans syndrome (BOS). OB is thought to result from chronic rejection leading to obliteration and scarring of the terminal bronchioles which causes a significant reduction in pulmonary function parameters, most specifically the forced expiratory volume in 1 second (FEV1). In the absence of confounding variables, lung transplant recipients are considered to suffer from BOS grade ≥1 if they experience a sustained (>3 weeks) ≥ 20% decline in FEV1 from a baseline of the average of the two best FEV1 measurements obtained at least 3 weeks apart.

Most immunosuppressive regimens after lung transplantation are based on calcineurin inhibitors. The introduction of cyclosporine was responsible for the initial success of lung transplantation in the early 1980s as it allowed the use of a lower dose of corticosteroids and hence afforded superior wound healing. Its chief mechanism of action is the blockade of T-lymphocyte activation by inhibiting interleukin-2 (IL 2) synthesis. Tacrolimus is a macrolide lactone that was introduced in the 1990s and is now widely accepted as an alternative to cyclosporine. Mechanisms of action and toxicities of tacrolimus and cyclosporine are similar, and tacrolimus has proven to be at least as effective as cyclosporine in solid organ transplantation including lung transplantation. Tacrolimus is approximately 50 times more potent than cyclosporine and has proven to be an effective rescue agent for patients with either recurrent or refractory acute allograft rejection. Whether denovo tacrolimus use can reduce the incidence of BOS when compared with cyclosporine after lung transplantation remains unclear. To date there are no published adequately powered randomized controlled trials in lung transplantation which compare the efficacy and safety of the calcineurin inhibitors cyclosporine and tacrolimus for primary immunosuppression.

The investigators therefore conducted a randomized, open-label, multi-center, investigator driven trial comparing tacrolimus with cyclosporine - both arms in combination with mycophenolate mofetil (MMF) and prednisolone for the prevention of BOS in lung and heart-lung transplant recipients.

The investigators chose to partner the calcineurin inhibitor with MMF instead of azathioprine. MMF is an ester prodrug of mycophenolic acid (MPA), a potent and specific inhibitor of de novo purine synthesis which blocks the proliferation of both T and B lymphocytes. The potential superiority of MMF over its comparator azathioprine after lung transplantation has been suggested in small and nonrandomized studies. However, large randomized trials in renal and heart transplantation have demonstrated the greater efficacy of MMF for preventing acute allograft rejection when compared with azathioprine.

The study protocol was accepted by each local hospital research ethics committee. All patients provided written informed consent and were free to withdraw from the study at any time point. The trial was proposed and designed by a steering committee consisting of members of the study group, The European and Australian Investigators in Lung Transplantation (EAILTx), representing experienced lung transplant centers from Australia, Austria, Belgium, Germany, Spain and Switzerland.

The study took place at 14 experienced lung transplantation centers in 5 European countries (Austria, Belgium, Germany, Spain and Switzerland) and Australia (Appendix). Patients were screened for eligibility prior to transplantation. At the time of transplantation, randomization was performed using a centralized telephone based computer randomization tool. Patients were assigned to receive tacrolimus, MMF and corticosteroids or cyclosporine, MMF and corticosteroids and were stratified according to whether they had cystic fibrosis (CF) or not. Stratification was performed because chronic airway infection, multi-organ involvement and variable gastrointestinal absorption pose specific clinical problems in individuals with CF which may have introduced an outcome bias if there were an imbalance of CF patients between groups.

Patients were followed for 3 years. Regular visits after transplantation were scheduled at 1 and 2 weeks, at 1, 2, 3, 6, 9, and 12 months, and every 6 months thereafter. Data were entered into an electronic case report form (eCRF) and regularly monitored and checked for inconsistencies by an independent monitor who was also responsible for query management. After completion of the follow-up period source data verification was performed by independent data management specialists who visited the centers and checked patient records for completeness of data.

The study was planned and designed in 1999, the protocol written in 2000, and the first patient randomized in 2001 at which time the registration of randomized trials was not mandatory. Reporting follows the Consort statement.

From January 2001 until June 2003 a total of 265 patients from 14 centers in 6 countries were randomized and transplanted.

ELIGIBILITY:
Inclusion Criteria:

* male or female recipients of a first heart-lung
* bilateral or single lung allograft suitable to receive triple immunosuppressive therapy with tacrolimus or cyclosporine, MMF and corticosteroids per standard guidelines
* Age range = 18-66 years
* Able to understand the purposes and risks of the study
* Female patients of child bearing age agreeing to maintain effective birth control practice during the follow-up period

Exclusion Criteria:

* need for immunosuppressive regimen other than study medication or received additional organ transplantations
* Pregnant women, nursing mothers or women unwilling to use adequate contraception
* Serologic evidence of human immunodeficiency virus, hepatitis B surface antigen or hepatitis C virus antibodies
* Panresistant infections with Burkholderia cepacia or mycobacteria during the last 12 months preceding lung transplantation
* Patients with renal insufficiency (creatinine clearance < 40 ml/min
* Patients in need of invasive ventilator devices or extracorporeal membrane oxygenation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2001-01; Primary Completion 2007-10 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence of bronchiolitis obliterans syndrome | 3 years post transplant
  The incidence of patients with bronchiolitis obliterans syndrome (BOS), defined as a sustained fall (for >1 month) in maximum FEV1 of 20% or more (compared to baseline) over three years post transplant.

SECONDARY OUTCOMES:
Acute allograft rejection | 3 years post transplant
  One- and 3-year rates of acute allograft rejection determined by clinical criteria or transbronchial lung biopsy.
Patient and graft survival | 3 years post transplant
  Patient and graft survival at one and three years
Incidence and spectrum of infections | 3 years post transplant
  Incidence and spectrum (viral, bacterial, fungal)of infections after transplantation
Renal failure | 3 years post transplant
  Post operative onset of renal dysfunction (defined as a persistent increase in serum creatinine of > 2mg/dl) or dialysis dependency
Treatment failure | 3 years post transplant
  Treatment failure defined as drug discontinuation (e.g. conversion to a different immunosuppression regimen)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Reichenspurner, MD, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany; Allan Glanville, MD, PhD, Study Chair — St Vincent's Hospital - Sydney, Australia; Hendrik Treede, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
Locations (14):
- St. Vincent's Hospital, Sydney, Australia
- Allgemeines Krankenhaus Wien, Vienna, Austria
- Belgium (2):
  - Hospital Erasme, Brussels
  - Universitaire Ziekenhuizen, Leuven
- Germany (4):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Kiel, Kiel
- Spain (5):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Clínica Puerta de Hierro, Madrid
  - Hospital Marques de Valdecilla, Santander
- Centre hospitalier universitaire vaudois, Lausanne, Switzerland

REFERENCES:
- [Background] Aurora P, Edwards LB, Kucheryavaya AY, Christie JD, Dobbels F, Kirk R, Rahmel AO, Stehlik J, Hertz MI. The Registry of the International Society for Heart and Lung Transplantation: thirteenth official pediatric lung and heart-lung transplantation report--2010. J Heart Lung Transplant. 2010 Oct;29(10):1129-41. doi: 10.1016/j.healun.2010.08.008. No abstract available. PMID 20870167
- [Background] Reichenspurner H, Girgis RE, Robbins RC, Conte JV, Nair RV, Valentine V, Berry GJ, Morris RE, Theodore J, Reitz BA. Obliterative bronchiolitis after lung and heart-lung transplantation. Ann Thorac Surg. 1995 Dec;60(6):1845-53. doi: 10.1016/0003-4975(95)00776-8. PMID 8787504
- [Background] Snell GI, Boehler A, Glanville AR, McNeil K, Scott JP, Studer SM, Wallwork J, Westall G, Zamora MR, Stewart S. Eleven years on: a clinical update of key areas of the 1996 lung allograft rejection working formulation. J Heart Lung Transplant. 2007 May;26(5):423-30. doi: 10.1016/j.healun.2007.01.040. No abstract available. PMID 17449409
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517
- [Background] Hachem RR, Yusen RD, Chakinala MM, Meyers BF, Lynch JP, Aloush AA, Patterson GA, Trulock EP. A randomized controlled trial of tacrolimus versus cyclosporine after lung transplantation. J Heart Lung Transplant. 2007 Oct;26(10):1012-8. doi: 10.1016/j.healun.2007.07.027. PMID 17919621
- [Background] Keenan RJ, Konishi H, Kawai A, Paradis IL, Nunley DR, Iacono AT, Hardesty RL, Weyant RJ, Griffith BP. Clinical trial of tacrolimus versus cyclosporine in lung transplantation. Ann Thorac Surg. 1995 Sep;60(3):580-4; discussion 584-5. doi: 10.1016/0003-4975(95)00407-C. PMID 7545889
- [Background] Treede H, Klepetko W, Reichenspurner H, Zuckermann A, Meiser B, Birsan T, Wisser W, Reichert B; Munich and Vienna Lung Transplant Group. Tacrolimus versus cyclosporine after lung transplantation: a prospective, open, randomized two-center trial comparing two different immunosuppressive protocols. J Heart Lung Transplant. 2001 May;20(5):511-7. doi: 10.1016/s1053-2498(01)00244-3. PMID 11343977
- [Background] Zuckermann A, Reichenspurner H, Birsan T, Treede H, Deviatko E, Reichart B, Klepetko W. Cyclosporine A versus tacrolimus in combination with mycophenolate mofetil and steroids as primary immunosuppression after lung transplantation: one-year results of a 2-center prospective randomized trial. J Thorac Cardiovasc Surg. 2003 Apr;125(4):891-900. doi: 10.1067/mtc.2003.71. PMID 12698153
- [Background] Sarahrudi K, Estenne M, Corris P, Niedermayer J, Knoop C, Glanville A, Chaparro C, Verleden G, Gerbase MW, Venuta F, Bottcher H, Aubert JD, Levvey B, Reichenspurner H, Auterith A, Klepetko W. International experience with conversion from cyclosporine to tacrolimus for acute and chronic lung allograft rejection. J Thorac Cardiovasc Surg. 2004 Apr;127(4):1126-32. doi: 10.1016/j.jtcvs.2003.11.009. PMID 15052212
- [Background] Vitulo P, Oggionni T, Cascina A, Arbustini E, D'Armini AM, Rinaldi M, Meloni F, Rossi A, Vigano M. Efficacy of tacrolimus rescue therapy in refractory acute rejection after lung transplantation. J Heart Lung Transplant. 2002 Apr;21(4):435-9. doi: 10.1016/s1053-2498(01)00379-5. PMID 11927219
- [Background] McNeil K, Glanville AR, Wahlers T, Knoop C, Speich R, Mamelok RD, Maurer J, Ives J, Corris PA. Comparison of mycophenolate mofetil and azathioprine for prevention of bronchiolitis obliterans syndrome in de novo lung transplant recipients. Transplantation. 2006 Apr 15;81(7):998-1003. doi: 10.1097/01.tp.0000202755.33883.61. PMID 16612275
- [Background] Orens JB, Estenne M, Arcasoy S, Conte JV, Corris P, Egan JJ, Egan T, Keshavjee S, Knoop C, Kotloff R, Martinez FJ, Nathan S, Palmer S, Patterson A, Singer L, Snell G, Studer S, Vachiery JL, Glanville AR; Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. International guidelines for the selection of lung transplant candidates: 2006 update--a consensus report from the Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2006 Jul;25(7):745-55. doi: 10.1016/j.healun.2006.03.011. No abstract available. PMID 16818116
- [Background] Shyu S, Dew MA, Pilewski JM, DeVito Dabbs AJ, Zaldonis DB, Studer SM, Crespo MM, Toyoda Y, Bermudez CA, McCurry KR. Five-year outcomes with alemtuzumab induction after lung transplantation. J Heart Lung Transplant. 2011 Jul;30(7):743-54. doi: 10.1016/j.healun.2011.01.714. Epub 2011 Mar 21. PMID 21420318
- See also: International Society For Heart and Lung Transplantation — http://www.ishlt.org/